CLINICAL TRIAL: NCT05313893
Title: A Clinical Trial to Assess Immunogencity and Safety of 2 Doses of anInactivated Quadrivalent Influenza Vaccine in Chinese Children Aged 3 to 8Years
Brief Title: A Clinical Trial of an Inactivated Quadrivalent Influenza Vaccine in Chinese Children Aged 3 to 8 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SJLGYM-2021-Ⅳ-01
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Safety; Immunogenicity; Quadrivalent influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects received 2 doses of an inactivated quadrivalent influenza vaccine,4 weeks apart. Blood samples were obtained from children at 3 time points-before receipt of dose 1, 4 weeks after receipt of dose 1 and before dose 2, and4 weeks after dose 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadrivalent influenza vaccine (Experimental): Subjects received 2 doses of 0.5 mL of quadrivalentinfluenza vaccine, 4 weeks apart. Each 0.5-ml dosecontained 15 μg of hemagglutinin per strain.
  Interventions: Biological: Quadrivalent influenza vaccine

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — Subjects receive two doses of quadrivalent influenzavaccine administered 4 weeks apart by intramuscularinjection. Each 0.5-ml dosecontained 15 μg of hemagglutinin per strain.

SUMMARY:
Routine annual influenza vaccination is recommended for all persons aged≥6 months who do not have contraindications. For those aged 6 monthsthrough 8 years who have previously received ≥2 total doses of trivalent orquadrivalent influenza vaccine ≥4 weeks apart, they require only 1 dose ofinfluenza vaccine. For those who have not previously received ≥2 doses oftrivalent or quadrivalent influenza vaccine, they require 2 dose of influenzavaccine. but the evidence on how to select vaccine doses for quadrivalentinfluenza vaccine is limited in China. The study is a prospective, open-labelcomparison of the immunogenicity and reactogenicity of 1 versus 2 doses ofan inactivated quadrivalent influenza vaccine in subjects of 3-8 years old withdifferent history of influenza vaccination.

DETAILED DESCRIPTION:
Subjects receive 2 dosed of quadrivalent influenza vaccine 4 weeks apart.Blood samples were obtained from children at 3 time points-before receiptof dose 1, 4 weeks after receipt of dose 1 and before dose 2, and 4 weeksafter dose 2. Hemagglutination inhibition (HAI) antibody titers to the A/H3N2,A/H1N1, and B antigens included in the vaccine were measured at each timepoint

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-8 years old
* Healthy subjects judged from medical history and clinical examination
* Subjects themselves or their guardians able to understand and sign theinformed consent
* Subjects themselves or their guardians can and will comply with therequirements of the protocol
* Subjects have received ≥2 doses of trivalent or quadrivalent infuenzavaccine before enrollment (Doses need not have been received duringsame or consecutive seasons); Subjects have not received infuenzavaccine before enrollment
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Any prior administration of other research medicine/vaccine in last 30 days
* Any prior administration of influenza vaccine in last 6 month
* Any prior administration of immunodepressant or corticosteroids in last 3 months
* Any prior administration of blood products in last 3 months
* Any prior administration of any attenuated live vaccine in last 14 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Subject who developed guillain-Barre syndrome post influenza vaccination
* Subject who is allergic to any ingredient of the vaccine
* Subject with acute febrile illness or infectious disease
* Thrombocytopenia, blood coagulation disorder or bleeding difficulties withintramuscular injection
* Subject with damaged or low immune function which has already beenknown
* Subject with congenital heart disease or other birth defects unsuitable for vaccination.
* Subject with respiratory diseases (including pneumonia, tuberculosis, severe asthma, etc.), heart, liver and kidney diseases, mental disorders, or chronic infections.
* Any medical, psychological, social or other condition judged byinvestigator, that may interfere subject's compliance with the protocol

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
the 95% confidence interval (CI) lower limit for Seroconversion Rate (SCR) of Hemagglutination inhibition (HAI)antibodies against each virus strain after 2nd vaccination ≥40% | day 28 after dose 2
  The lowest dilution used in the assay is 1/10. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥ four-fold increase in post-vaccination titer.
Number of participants with Adverse Reactions (ARs) | 28 days after each vaccination
  Frequency and severity of ARs for 28 days after each vaccination

SECONDARY OUTCOMES:
the 95% CI lower limit for seroprotection rates of HAI antibodies against each virus strain after 2nd vaccination≥70% | day 28 after dose 2
  A seroprotected subject is defined as a vaccinated subject with serum HAI titer≥ 1:40.
Geometric Mean Fold Increase (GMFI) of HAI titer against each virus strain after 2nd vaccination>2.5 | day 28 after dose 2
  Hemagglutination inhibition (HAI) titers were used to calculate post-vaccination geometric mean fold increase (GMFI)against each virus strain
Number of participants with Adverse Events (AEs) | 28 days after each vaccination
  Frequency and severity of AEs for 28 days after each vaccination
Number of participants with Serious Adverse Events (SAE) | 6 months after the last vaccination
  Frequency of SAEs for 6 months after the last vaccination

OTHER OUTCOMES:
Comparision between Seroconversion Rate (SCR) of HAI antibodies against each virus strain post dose 1 and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2
  The lowest dilution used in the assay is 1/10. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥ four-fold increase in post-vaccination titer.
Comparision between Geometric Mean Titre (GMT) of HAI antibodies against each virus strain post dose 1 and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2
Comparision between seroprotection rates of HAI antibodies against each virus strain post dose 1 and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2
  A seroprotected subject is defined as a vaccinated subject with serum HAI titer≥ 1:40.
Comparision between Geometric Mean Fold Increase (GMFI) of HAI antibodies against each virus strain post dose 1and dose 2 | day 28 after receipt of dose 1 and before dose 2, and day 28 after dose 2

CONTACTS AND LOCATIONS:
Locations (1):
- Donghai County Center for Disease Control and Prevention, Lianyungang, Jiangsu, China